CLINICAL TRIAL: NCT05347966
Title: The Canadian Therapeutic Platform Trial for Multidomain Interventions to Prevent Dementia: Brain Health Support Program Intervention
Brief Title: Brain Health Support Program
Acronym: CTU: BHSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CTU: BHSP
Record Dates: First submitted 2022-04-14; First posted 2022-04-27 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Dementia Prevention; Mild Cognitive Impairment; Subjective Cognitive Impairment; Cognitive Change
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain Health PRO (Other)
  Interventions: Other: Brain Health PRO

INTERVENTIONS:
Other: Brain Health PRO — BHPro is a 45-week, multidomain web-based formal educational program which has been designed to increase dementia literacy, convey best available evidence for lifestyle changes that can mitigate dementia risk, and foster engagement toward one's own brain health.
  Other Names: BHPro

SUMMARY:
The Canadian Therapeutic Platform Trial for Multidomain Interventions to Prevent Dementia (CAN-THUMBS UP, or CTU) is a comprehensive and innovative program aimed to develop, implement and evaluate an interactive and compelling online educational Brain Health Support Program (BHSP) intervention, called Brain Health PRO (BHPro), with potential to positively influence dementia literacy, lifestyle risk factors, and scale-up to reach the broader Canadian public; enroll and retain a community-dwelling Platform Trial Cohort (PTC) of individuals at risk of dementia; and support an open platform trial to test a variety of multidomain interventions that might further benefit individuals at risk of dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Completion and documentation of the electronic Informed Consent Process (from the participant)
2. Sufficient proficiency in English or French to undergo remote clinical and neuropsychological assessment and participate in an online educational program.
3. Technical ability to participate in an online educational program and remote assessments (i.e. computer and internet access; ability to send and receive emails; ability to complete remote assessments)
4. Sufficient vision and hearing to participate in online educational program and to undergo remote clinical and neuropsychological testing
5. Ability to sit comfortably for a period of about 30 minutes
6. Ages 60-85
7. Meets criteria for No Dementia and meet criteria [according to Canadian Consortium on Neurodegeneration in Aging (CCNA) Criteria, Appendix 1] of one of the following:

   * Cognitively Unimpaired (CU)
   * Cognitively Unimpaired plus Subjective Cognitive Impairment (CU + SCI)
   * Mild Cognitive Impairment (MCI)
8. AND Classified as being at increased risk of dementia based on at least one of the following:

   * First-degree family history of dementia
   * Self-Reported or documented current and/or history at midlife (45-60 years) on any of the following lifestyle risk factors:

   Hypertension (documented Systolic Blood Pressure > 140 mm Hg; OR physician diagnosis of hypertension; OR treatment for hypertension; OR other approaches to treatment (e.g. diet, exercise)) Hypercholesterolemia (documented total cholesterol > 6.5 mmol/L; OR physician diagnosis of hypercholesterolemia; OR treatment for hypercholesterolemia; OR other approaches to treatment (e.g. diet, exercise) Body Mass Index > 30 kg/m2 (derived from NIH Metric BMI Calculator) Physical Inactivity (active is defined as engaging in a minimum of 20- 30 min of physical activity causing sweating and breathlessness, at least 2 times a week)
9. Participant has a family physician or other healthcare provider and agrees to have the provider notified of participation in the study and incidental or other findings that may be clinically significant

Exclusion Criteria:

1. Participants who, in the opinion of the investigator, are not able to complete trial procedures remotely or adhere to the schedule of study assessments will be excluded from study participation.
2. Individuals where English or French is not sufficiently proficient for remote clinical assessment, neuropsychological testing and participation in an online educational program.
3. Participants who do not have sufficient vision and hearing for remote clinical assessment, neuropsychological testing participation in an online educational program
4. Individuals who do not have the technical ability to participate in an online educational program. Technical ability is defined as having computer and internet access; ability to send and receive emails; ability to participate in remote assessments
5. Individuals who have a clinical diagnosis of Dementia
6. Clinical Dementia Rating (CDR; telephone/video-conference administration) Score of >1
7. Total Score on the Montreal Cognitive Assessment (MoCA; video-conference administration) <13

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - University of British Columbia, Vancouver, British Columbia
  - University of New Brunswick, Fredericton, New Brunswick
  - Cape Breton University, Cape Breton, Nova Scotia
  - Cognitive Clinical Research Group, Parkwood Research Institute, London, Ontario
  - Gait and Brain Laboratory, Parkwood Research Institute, London, Ontario
  - Baycrest, Toronto, Ontario
  - CRIUGM/ CIUSSS du Centre-Sud-de-l'Île-de-Montréal, Montreal, Quebec

REFERENCES:
- [Derived] Belleville S, Anderson ND, Bherer L, Camicioli R, Carrier J, Chan S, Cuesta M, Dang-Vu TT, Dwosh E, Fiocco AJ, Ferland G, Gilbert B, Harris E, Itzhak I, Jarrett P, Kadri MA, Laurin D, Liu-Ambrose T, McGibbon CA, Middleton L, Miller L, Nygaard HB, Montero-Odasso M, Murphy K, Phillips N, Pichora-Fuller MK, Robillard JM, Smith EE, Speechley M, Trigui A, Wittich W, Chertkow H, Feldman HH; CTU expert group for the Canadian Consortium on Neurodegeneration in Aging (CCNA), CAN-THUMBS UP Study Group. Brain health PRO/Sante cerveau PRO: The development of a web-based program for dementia literacy and risk factor reduction. J Prev Alzheimers Dis. 2025 Jun;12(6):100134. doi: 10.1016/j.tjpad.2025.100134. Epub 2025 Mar 15. PMID 40090784
- [Derived] Feldman HH, Belleville S, Nygaard HB, Montero-Odasso M, Durant J, Lupo JL, Revta C, Chan S, Cuesta M, Slack PJ, Winer S, Brewster PWH, Hofer SM, Lim A, Centen A, Jacobs DM, Anderson ND, Walker JD, Speechley MR, Zou GY, Chertkow H. Protocol for the Brain Health Support Program Study of the Canadian Therapeutic Platform Trial for Multidomain Interventions to Prevent Dementia (CAN-THUMBS UP): A Prospective 12-Month Intervention Study. J Prev Alzheimers Dis. 2023;10(4):875-885. doi: 10.14283/jpad.2023.65. PMID 37874110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged 60-85 who were cognitively unimpaired, or had subjective cognitive impairment, or mild cognitive impairment, and at least one pre-defined risk factor for dementia, among other specific criteria, were eligible to participate in this study. A total of 354 participants were enrolled at 7 centres across Canada. Recruitment began in April 2022 and the last participant exited the study in April 2024.
Pre-assignment Details: Participants who did not meet eligibility criteria for the study screen-failed before the baseline visit.
Groups:
- BHSP-Main: Brain Health PRO (BHPro) is an innovative online platform designed to help reduce the risk of dementia by providing individuals with the tools and knowledge needed to make positive lifestyle changes. The program offers a flexible, user-friendly interface that allows users to assess their risk and engage with educational modules specifically tailored to their needs.
Period: Overall Study
Arm/Group | BHSP-Main
Started | 354
Completed | 315
Not Completed | 39

BASELINE CHARACTERISTICS:
Population: A total of 354 participants were eligible for the study with one participant requesting their data not be used, leaving 353 baseline participants to report on.
Groups:
- BHSP Main: Brain Health PRO (BHPro) is an innovative online platform designed to help reduce the risk of dementia by providing individuals with the tools and knowledge needed to make positive lifestyle changes. The program offers a flexible, user-friendly interface that allows users to assess their risk and engage with educational modules specifically tailored to their needs.
Arm/Group | BHSP Main
Number analyzed (Participants) | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245
  Male | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 352
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 318
  Asian | 12
  Multiple Ethnicities | 8
  Other | 15
Region of Enrollment [Number; unit: participants]
  Canada | 353

OUTCOME MEASURES:

1. Primary Outcome: Change in Dementia Literacy From Baseline to Month 12
Description: The primary outcome will be change in dementia literacy following participation in the study, as measured by the Alzheimer's Disease Knowledge Scale (ADKS). The ADKS is designed to assess knowledge about Alzheimer's Disease (AD) among laypeople, patients, caregivers, and professionals. This self-report questionnaire contains 30 true/false items. The total score is the sum of the scores from the 30 items, which is quantitative and ranges from 0-30, with a higher score indicating better knowledge about AD. To aide interpretation, change in ADKS scores were converted to standardized change scores by dividing the covariate-adjusted least squares mean change by the baseline standard deviation. The results reported are the standardized change on the scale from baseline to month 12. The converted to standardized score range is -10.81 to +10.81. The greater the positive change in score, the greater the increase in knowledge of dementia.
Time Frame: 12 months
Population: Intention To Treat (ITT) sample: Includes all participants who (1) meet screening criteria (2) and completed at least 1 assessment at baseline. Covariates include: age, sex, race, cognitive status, and Heaton education score.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | BHSP Main
Number analyzed (Participants) | 353
Score on a scale | 0.191 [-0.014 to 0.397]

2. Secondary Outcome: Change in Self-efficacy From Baseline to Month 12
Description: Change in self-efficacy following participation in the study, as measured by the General Self-Efficacy Scale (GSE). The GSE measures perceived competence in dealing with a range of stressful or challenging situations. This self-report questionnaire contains 10-items, each rated on a 4-point scale (not true at all, hardly true, moderately true, exactly true). The total score is the sum of the scores for the 10 items, which is quantitative and ranges from 10-40, with a higher score indicating more self-efficacy. To aide interpretation, change in GSE scores were converted to standardized change scores by dividing the covariate-adjusted least squares mean change by the standard deviation. The results reported are the standardized change on the scale from baseline to month 12. The converted to standardized score range is -7.39 to +7.39. The greater the change in score, the greater the increase in self-efficacy.
Time Frame: 12 months
Population: Intention to Treat sample (ITT) sample: includes all participants who (1) meet screening criteria (2) and completed at least 1 assessment at baseline. Covariates include: age, sex, race, cognitive status, and Heaton education score
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BHSP Main
Number analyzed (Participants) | 353
score on a scale | 0.157 [0.042 to 0.272]

3. Secondary Outcome: To Evaluate Usability of BHPro
Description: Based on System Usability Scale (SUS). The SUS is an 11-item questionnaire with 5-point Likert scale. The total raw score ranges from 0-43 with a higher score indicating greater usability and satisfaction with Brain Health Pro.
Time Frame: 12 months
Population: 248 of 353 participants completed the System Usability Scale at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BHSP Main
Number analyzed (Participants) | 248
score on a scale | 34 (6)

4. Secondary Outcome: Number of Chapters Completed on BHPro
Description: To evaluate engagement with Brain Health PRO, the number of chapters completed on BHPro was calculated. There is a total of 180 chapters (181 when orientation chapter is included) that are available on BHPro. The program allows participants to view 160 chapters (excluding the orientation chapter) when reaching week 45 (the intended length of the BHPro program). After 45 weeks, the remaining chapters that were still locked will become accessible for users interested in viewing all the program content. The range of chapters that could be completed on Brain Health PRo by participants is 1-181, with a higher number indicating higher engagement with the program.
Time Frame: 12 months
Population: Modified Intention To Treat (mITT) sample: Includes all eligible participants who (1) have completed at least one assessment for the outcome of interest and (2) registered for BHPro.
Measure: Mean (Standard Deviation); unit: Chapters completed
Arm/Group | BHSP Main
Number analyzed (Participants) | 345
Chapters completed | 142 (60)

5. Secondary Outcome: To Evaluate User Acceptance of BHPro With the Technology Acceptance Model Questionnaire (TAMQ).
Description: Based on Technology Acceptance Model Questionnaire. The TAMQ is a 20-item questionnaire (adapted for BHPro) with 7-point scale. The total score ranges between 0-120, with a higher score indicating greater acceptance and satisfaction with BHPro.
Time Frame: 12 months
Population: 257 of 353 participants completed the Technology Acceptance Model Questionnaire at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BHSP Main
Number analyzed (Participants) | 257
score on a scale | 94 (18)

ADVERSE EVENTS:
Time Frame: Adverse event data is collected from Baseline up to 30 days after study participation has ended. This is approximately 1 year for participants who remained in the study until the end and less time for those who withdrew early. Systematic collection of AEs occurred at the following study visits: Baseline, Month 6, Month 12. Non-systematic AE reporting, spontaneous reporting by participant, was also implemented.
Description: The study protocol defines an adverse event (AE) as any unfavourable or unintended sign, symptom, or disease associated with study procedures that are both non-serious and either temporally or causally related to study procedures. To be reported as a Serious Adverse Event (SAE), the protocol requires that the event must be serious, unanticipated, and related to study procedures. All-cause mortality, SAEs, and Other (Not Including Serious) AEs not related to study procedures were not collected.
Arm/Group | BHSP Main
All-Cause Mortality (participants affected / at risk) | 0/353
Serious Adverse Events (participants affected / at risk) | 0/353
Other Adverse Events (participants affected / at risk) | 3/353
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BHSP Main (N=353)
Skin Reaction likely related to EEG headband (Skin and subcutaneous tissue disorders) | 2 (2)
Headache likely related to EEG headband (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT05347966/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT05347966/SAP_001.pdf